CLINICAL TRIAL: NCT06647745
Title: A Randomized, Double-blind, Multi-center, Active-controlled, Phase 3 Clinical Trial to Evaluate the Efficacy and Safety of Combination Therapy of THP-00101, THP-00102, and THP-00103 in Subjects With T2DM and Essential Hypertension
Acronym: THP-001-031
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: THPharm Corp. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: THP-001-031
Record Dates: First submitted 2024-10-16; First posted 2024-10-18 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Type 2 Diabetes; Hypertension
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension | interventions — dapagliflozin; Telmisartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Study group (Experimental): The participant will receive the investigational drugs THP-00101 (Dapagliflozin 10 mg), THP-00102 (Telmisartan 80 mg), and a placebo for THP-00103 once a day by per oral over 12 weeks
  Interventions: Drug: THP-00101; Drug: THP-00102; Drug: THP-00106
- Control group 1 (Placebo Comparator): The participant will receive the investigational drugs THP-00101 (Dapagliflozin 10 mg), Placebo of THP-00102, and Placebo of THP-00103 once a day by per oral over 12 weeks
  Interventions: Drug: THP-00101; Drug: THP-00104; Drug: THP-00105
- Control group 2 (Placebo Comparator): The participant will receive the investigational drugs Placebo of THP-00101, THP-00102 (Telmisartan 80 mg), and Placebo of THP-00103 once a day by per oral over 12 weeks
  Interventions: Drug: THP-00102; Drug: THP-00104; Drug: THP-00106
- Exploratory group (Other): The participant will receive the investigational drugs THP-00101 (Dapagliflozin 10 mg), Placebo of THP-00102, and THP-00103 (Telmisartan 40 mg) once a day by per oral over 12 weeks
  Interventions: Drug: THP-00101; Drug: THP-00103; Drug: THP-00105

INTERVENTIONS:
Drug: THP-00101 — Dapagliflozin 10 mg
  Other Names: Forxiga Tab. 10mg
  Arms: Control group 1; Exploratory group; Study group
Drug: THP-00102 — Telmisartan 80 mg
  Other Names: Micardis Tab. 80mg
  Arms: Control group 2; Study group
Drug: THP-00103 — Telmisartan 40 mg
  Other Names: Micardis Tab. 40mg
  Arms: Exploratory group
Drug: THP-00104 — Placebo of Dapagliflozin 10mg
  Other Names: Placebo of Fociga Tab. 10mg
  Arms: Control group 1; Control group 2
Drug: THP-00105 — Placebo of Telmisartan 80mg
  Other Names: Placebo of Micardis Tab. 80mg
  Arms: Control group 1; Exploratory group
Drug: THP-00106 — Placebo of Telmisartan 40mg
  Other Names: Placebo of Micardis Tab. 40mg
  Arms: Control group 2; Study group

SUMMARY:
[Primary Objective] To demonstrate the superiority of the change in mean sitting systolic blood pressure (MSSBP) and hemoglobin A1c (HbA1c)on week 12 of the combination therapy of THP-00101 (dapagliflozin 10 mg) and THP-00102 (telmisartan 80 mg) compared to THP-00101 or THP-00102 monotherapy among subjects with type 2 diabetes mellitus accompanied by essential hypertension. [Secondary Objective] To comparatively evaluate secondary efficacy and safety in the THP-00101 monotherapy group, THP-00102 monotherapy group, THP-00101 and THP-00102 combination therapy group, and THP-00101 and THP-00103 (telmisartan 40 mg) combination therapy group among subjects with type 2 diabetes mellitus accompanied by essential hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Screening (V1)

  1. Adult males and females aged 19 (the legal adult age of each country) and above on the date of written informed consent
  2. Subjects with type 2 diabetes mellitus accompanied by essential hypertension
  3. Subjects with the following hemoglobin A1c (HbA1c) and fasting plasma glucose (FPG) levels at screening (V1)*
* hemoglobin A1c less than or equal to 9.5% and more than 6.5%
* fasting plasma glucose less than or equal to 270 mg/dL

  * Including subjects who did not use oral hypoglycemic agents within 8 weeks from screening and subjects who took metformin monotherapy or dual combination therapy that included metformin for 8 weeks or longer from screening 4. Subjects with the following mean sitting systolic blood pressure (MSSBP) measured in the reference arm** at screening (V1)***
* If not taking antihypertensive agents: MSSBP less than 160 mmHg and more than 140 mmHg
* If taking antihypertensive agents: MSSBP less than 160 mmHg and more than 130 mmHg **Reference arm: The arm with the higher MSSBP after measuring it 3 times in each arm at screening (V1) (If the MSSBP is the same between both arms, then the arm with the higher mean sitting diastolic blood pressure (MSDBP) is selected as the reference arm.)

  ***Classified based on whether antihypertensive agents were administered within 4 weeks from screening (V1) 5 Subjects considered by the investigator appropriate to discontinue the use of oral hypoglycemic agents and antihypertensive agents, other than the existing metformin, during the study (with metformin maintained at a minimum of 1,000 mg/day) 6 Subjects who received a sufficient explanation of the objectives and content of the study and voluntarily provided written informed consent
* Baseline (V2)

  1. Subjects with the following HbA1c and FPG levels at baseline (V2) - HbA1c less than or equal to 9.5% and more than 6.5% - FPG less than or equal to 270 mg/dL 2. Subjects with the following MSSBP measured in the reference arm at baseline (V2) - MSSBP less than 160 mmHg and more than 140 mmHg 3. Subjects who did not take oral hypoglycemic agents other than the same dose of metformin (More than 1,000 mg/day) for at least 8 weeks before baseline (V2) 4. Subjects who did not take antihypertensive agents for at least 2 weeks before baseline (V2) 5. Subjects with no disqualifying inclusion/exclusion criteria of screening (V1) when evaluating eligibility again at baseline (V2) 6. Subjects with compliance of 70% or higher with the investigational product during the run-in period
* Extension Period

  1. Subjects who have completed all procedures of the treatment period. Subjects who are unsuitable to participate in the study of the extension period, considering safety, etc., can be excluded.
  2. Subjects who received a sufficient explanation of the objectives and content of the extension period study and voluntarily provided written informed consent

     Exclusion Criteria:

  1. Subjects with the following blood pressures measured at screening (V1) and randomization (V2)

  (1) Subjects with the following MSDBP measured in the reference arm
* MSDBP ≥110 mmHg (2) Subjects with the following difference in mean blood pressure measured three times consecutively in each arm at least 2 minutes apart at screening (V1): MSSBP ≥20 mmHg and MSDBP ≥10 mmHg 2. Subjects with a BMI of >35 kg/m2 3. Subjects with the following comorbidities or conditions

  1. Mild to severe hepatic impairment
  2. Biliary obstruction or cholestasis
  3. AST or ALT ≥2 x ULN
  4. Total bilirubin >2 x ULN
  5. Patients with moderate (stage 3b) or severe renal impairment (eGFR by IDMS-MDRD <45 mL/min/1.73 m2)
  6. Acute conditions that may affect renal function, such as dehydration, severe infection, cardiovascular collapse (shock), and sepsis
  7. Diabetic precoma and coma
  8. Severe infection or severe traumatism
  9. Malnutrition, starvation, debilitation, pituitary insufficiency, or adrenal dysfunction
  10. Acute or chronic diseases that may cause tissue hypoxia such as respiratory failure (pulmonary infarction and severe pulmonary dysfunction) and shock, and gastrointestinal disorders including dehydration, diarrhea, and vomiting
  11. Orthostatic hypotension with symptoms
  12. Clinically significant ventricular tachycardia, atrial fibrillation, atrial flutter, or other arrhythmia considered clinically significant as judged by the investigator
  13. Hypertrophic obstructive cardiomyopathy, severe obstructive coronary artery disease, aortic stenosis, hemodynamically significant aortic valve or mitral valve stenosis
  14. Wasting diseases, autoimmune diseases, and connective tissue diseases
  15. Dysuria, anuria, oliguria, and ischuria that cannot be controlled by drugs
  16. Gastrointestinal diseases that may affect the absorption of the investigational product (gastrointestinal ulcer, gastritis, gastric spasm, gastroesophageal reflux disease, Crohn's disease, etc.)
  17. Subjects who are HBsAg positive§ or HCV antibody positive∥

      §Subjects who are taking antiviral products stably may participate

      ∥Subjects with negative HCV RNA test results may participate
  18. Subjects who are positive for HIV Ag/Ab combo test 4. Subjects with the following past medical history

  <!-- -->

  1. Hereditary angioedema or angioedema caused by ACE inhibitor or angiotensin II antagonist treatment.
  2. Hereditary problems such as galactose intolerance, Lapp lactose deficiency, glucose-galactose malabsorption, etc.
  3. Type 1 diabetes mellitus, secondary diabetes mellitus, lactic acidosis, acute or chronic metabolic acidosis, and ketoacidosis including diabetic ketoacidosis accompanied or not accompanied by coma
  4. Drug abuse or alcohol abuse
  5. Past medical history of secondary hypertension or all medical history suspected of secondary hypertension (not limited to the following: coarctation of aorta, primary hyperaldosteronism, renal artery stenosis, Cushing's syndrome, pheochromocytoma, polycystic kidney disease, etc.)
  6. Severe cardiac failure (NYHA class III and IV), ischemic heart disease (unstable angina and myocardial infarction), and peripheral vascular diseases that occurred within 24 weeks before screening (V1)
  7. Severe cerebrovascular diseases (stroke, cerebral infarction, cerebral hemorrhage, etc.) that occurred within 24 weeks before screening (V1)
  8. Moderate or malignant retinopathy that occurred within 24 weeks before screening (V1) (retinal hemorrhage, visual disturbance, and retinal microaneurysm that occurred within the last 24 weeks)
  9. Urinary tract infection or genital infection that occurred within 16 weeks before screening (V1)
  10. Malignant tumors that occurred within the last 5 years. Subjects who experienced no recurrence for at least 5 years after being declared cured or in the cases of basal cell carcinoma, squamous cell carcinoma of the skin, thyroid cancer, or carcinoma in situ at other sites, subjects who experienced no recurrence for at least 3 years after being declared cured can be enrolled based on the investigator's medical judgment 5. Subjects who received the following medication or non-pharmacological therapy at screening (V1)

  <!-- -->

  1. Bariatric surgery or lap-band surgery within 12 months before screening (V1)
  2. Percutaneous transluminal coronary angioplasty or coronary artery bypass graft surgery within 24 weeks before screening (V1)
  3. Antiobestic drugs or drugs based on the investigator's judgment to be capable of having significant effects on weight control within 12 weeks before screening (V1)
  4. Systemic corticosteroids used for 2 weeks or longer, within 8 weeks before screening (V1) (inhaled and topical agents, eye drops, intranasal, intra-articular administration, and other localized administrations are allowed regardless of duration)
  5. Insulin injections or GLP-1 receptor agonists administered for more than 7 days consecutively or non-consecutively within 8 weeks before screening (V1)
  6. Current treatment by the triple combination of antihypertensive agents, or current treatment by the dual combination including high-dose amlodipine (10 mg)
  7. Current treatment by the monotherapy of hypoglycemic agents except metfomin or current treatment by the triple combination including metformin
  8. Current treatment with drugs containing aliskiren
  9. Subjects currently receiving dialysis
  10. Scheduled tests involving the intravenous administration of radiographic iodinated contrast agents from 48 hours before the run-in period until the end of the study (e.g., intravenous urography, intravenous angiography, vascular angiography, computed tomography using contrast agents, etc.) 6. Subjects who are hypersensitive to the active ingredients (dapagliflozin or telmisartan) or other ingredients of the investigational product 7. Subjects with a history of hypersensitivity to metformin or biguanides 8. Subjects who participated in other clinical trials within 12 weeks before taking the investigational product of this study and were administered (or received) other investigational products (or devices) 9. Pregnant or breastfeeding women 10. Women and men of childbearing potential who have plans for pregnancy or do not agree to perform appropriate contraception from screening (V1) until 4 weeks after the last dose of the investigational product. The appropriate contraceptive methods for this study are as follows:

  <!-- -->

  1. Hormonal contraceptives (oral products, injections, implants, etc.)
  2. IUD or IUS
  3. Male or female sterilization (e.g., vasectomy, hysterectomy, bilateral oophorectomy, bilateral salpingectomy, etc.)
  4. Dual methods: Simultaneous use of 1) to 3) methods and the barrier method¶ or simultaneous use of double barrier methods# (simultaneous use of cap/diaphragm and male condom) and the spermicide
  5. Sexual abstinence: It is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatments. However, if the age, job, lifestyle, or sexual orientation of the participant assures contraception according to the investigator's decision, strict abstinence from sexual intercourse is also allowed. Periodic sexual abstinence (e.g., calendar method, symptothermal method, post-ovulation method, etc.) and withdrawal (coitus interruptus) are not acceptable methods of contraception.

     * Male condom, female condom, cap, diaphragm, sponge, etc. #However, simultaneous use of male condoms and female condoms is not allowed 11. Subjects unsuitable to participate in this study based on the investigator's judgment.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 221 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Changes in Hemoglobin A1c (HbA1c) | 12 weeks
  The Hemoglobin A1c will be measured using the high-performance liquid chromatography (HPLC) method.
Changes in Mean Sitting Systolic Blood Pressure (MSSBP) | 12 Weeks
  When using a digital blood pressure monitor, the subject should sit on a chair with their back supported, relax for at least 5 minutes, and keep their arm at heart level during the measurement

SECONDARY OUTCOMES:
Changes in glycemic parameter: hemoglobin A1c | 4, 8, and 12 weeks from baseline
  HbA1c will be measured
Changes in glycemic parameter: fasting plasma glucose | 4, 8, and 12 weeks from baseline
  FPG will be measured
Changes in glycemic parameter: homeostasis model assessment of insulin resistance (HOMA-IR) | 4, 8, and 12 weeks from baseline
  HOMA-IR will be measured using high-performance liquid chromatography and the hexokinase method.
Changes in glycemic parameter: homeostasis model assessment of beta-cell function (HOMA-beta) | 4, 8, and 12 weeks from baseline
  HOMA-beta will be measured using high-performance liquid chromatography and the hexokinase method
Changes in blood pressure: mean sitting systolic blood pressure | 4, 8, and 12 weeks from baseline
  When using a digital blood pressure monitor, the subject should sit on a chair with their back supported, relax for at least 5 minutes, and keep their arm at heart level during the measurement
Changes in blood pressure: mean sitting diastolic blood pressure | 4, 8, and 12 weeks from baseline
  When using a digital blood pressure monitor, the subject should sit on a chair with their back supported, relax for at least 5 minutes, and keep their arm at heart level during the measurement
Changes in blood pressure: pulse pressure | 4, 8, and 12 weeks from baseline
  When using a digital blood pressure monitor, the subject should sit on a chair with their back supported, relax for at least 5 minutes, and keep their arm at heart level during the measurement
Changes in blood pressure: percentage of normalized blood pressure | 4, 8, and 12 weeks from baseline
  When using a digital blood pressure monitor, the subject should sit on a chair with their back supported, relax for at least 5 minutes, and keep their arm at heart level during the measurement
Changes in blood pressure: response rate of blood pressure | 4, 8, and 12 weeks from baseline
  When using a digital blood pressure monitor, the subject should sit on a chair with their back supported, relax for at least 5 minutes, and keep their arm at heart level during the measurement

CONTACTS AND LOCATIONS:
Locations (2):
- The Catholic University of Korea, Yeouido ST. Mary's Hospital, Seoul, South Korea
- Thammasat University Hospital, Pathum Thani, Changwat Pathum Thani, Thailand

IPD SHARING:
Plan to Share IPD: Undecided